CLINICAL TRIAL: NCT04993573
Title: Acceptability, Representations and Experiences of the COVID-19 Pandemic : the ARECOVID Project
Brief Title: Acceptability, Representations and Experiences of the COVID-19 Pandemic
Acronym: ARECOVID
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Collaborators: Jean Monnet University (Other); Saint Etienne School of Mine (Other); Gerontopole Auvergne Rhone-Alpes (AURA) (Other)
Responsible Party: Sponsor
Other Study IDs: GA-2021-02
Record Dates: First submitted 2021-08-05; First posted 2021-08-06 (Actual); Last update posted 2021-08-06 (Actual); Status verified 2021-08

CONDITIONS: Aging
Keywords: COVID-19; caregivers; older; ageism; public health; hospital
MeSH Terms: conditions — COVID-19; Ageism | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Caregivers: Caregivers who work with older patients will be included. They will have a questionnaire
  Interventions: Other: Questionnaire
- Older: Older 65 people who live alone in their house will be included. They will have Individual interviews.
  Interventions: Other: Individual interview

INTERVENTIONS:
Other: Questionnaire — Questions about the impact of COVID-19 in their works
  Groups: Caregivers
Other: Individual interview — Discussion between the searcher and the participant about representations of COVID-19 and experiences about confinement.
  Groups: Older

SUMMARY:
The "ARECOVID" project is a comprehensive sociological study of what is being played out in organizational terms in the face of the COVID-19 pandemic. Through quantitative methods (questionnaires) and qualitative methods (semi-directive interviews), we would understand the essential views of the populations concerned by COVID-19, but also that of actors taking care of vulnerable elderly non-COVID. Special attention will be paid to the care pathway of elderly people with and without the virus, in a health system in full reorganization. We will try to understand the needs and experiences of all health actors (hospital/city) involved in COVID-19 and the experience of confinement and the Covid-19 of the elderly living at home, in order to reflect on a possible improvement in the health response of elderly people in the event of an epidemic health crisis.

DETAILED DESCRIPTION:
understand the needs and experiences of all health actors (hospital/city) involved in COVID-19 and the experience of confinement and the Covid-19 of the elderly living at home

ELIGIBILITY:
Inclusion Criteria:

* For older people : minimum age : 65 years
* For caregivers : works in gerontology

Exclusion Criteria:

* Person with a neurological disease
* Person under guardianship or curatorship

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Older 65 people Caregivers who works in gerontology
Sampling Method: Probability Sample
Enrollment: 520 (Actual)
Dates: Start 2020-07-01 (Actual); Primary Completion 2020-07-30 (Actual); Study Completion 2020-07-30 (Actual)

PRIMARY OUTCOMES:
Analysis representations of COVID-19 and confinement of older people | Day 20
  Measure by individual interviews

SECONDARY OUTCOMES:
Analysis impacts of COVID-19 in works of caregivers | Day 20
  Measure by questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Pauline Gouttefarde, Study Chair — Gerontopole Auvergne Rhone-Alpes (AURA)
Locations (1):
- Gérontopole AURA, Saint-Etienne, France